CLINICAL TRIAL: NCT02773953
Title: Impact of Telemonitoring on Delay of Intervention to Improve Precocious Adherence in CPAP-treated Sleep Apnea Patients
Brief Title: Impact of Telemonitoring to Improve Adherence in Continuous Positive Airway Pressure (CPAP)-Treated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK/16-03-39/4634
Record Dates: First submitted 2016-04-25; First posted 2016-05-16 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP; Telemonitoring
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP + T4PTelemonitoring device (Experimental): T4P® (Telemonitoring device) is added to CPAP at home. Sleep lab technical staff are connecting to the web portal 2 X/ week. In case of air leaks, persistant significant apnea-hypopnea index, use < 3h on three consecutive days, they have to call the patient .
  Interventions: Device: T4PTelemonitoring; Device: CPAP
- CPAP standard care (Active Comparator): After CPAP titration night, patients are instructed to use the device each night for the whole night. They receive written instruction and can reach the sleep unit (phone call, visit) how often they need, during week days, to resolve CPAP-related problems. A group educational session is scheduled 1 month after and a visit to the pneumologist 1.5 months after.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: T4PTelemonitoring — addition of a Telemonitoring unit on the CPAP line to standard care.
  Arms: CPAP + T4PTelemonitoring device
Device: CPAP — CPAP treatment for treatment of obstructive sleep apnea syndrome

SUMMARY:
Improvement in CPAP adherence can be obtained by usingTelemonitoring. T4P® is a telemonitoring unit added on CPAP device allowing to obtain a daily report of usage duration, mask leaks, pressure and apnea-hypopnea index. The purpose of this study is to assess the impact of telemonitoring on the delay to the first technical intervention after CPAP titration night in CPAP-treated obstructive sleep apnea patients managed in the sleep unit. The shortening of this delay could help to improve adherence during the first weeks of treatment. As a secondary aim, the investigators would like to assess the impact of telemonitoring on mean adherence during the first 3 months of treatment, which is a crucial period.

DETAILED DESCRIPTION:
Introduction CPAP (continuous positive airway pressure) is the most frequently used and effective treatment for obstructive sleep apnea syndrome (OSAS).

It has been proven to offer a survival benefit in patients with severe disease, to improve sleep quality, health-related quality of life and to decrease cardiovascular events, such as stroke and myocardial infarction.

The challenge of this treatment remains to obtain adequate adherence, defined as use during at least 4 hours/night and for more than 70% of the nights . Independently of this usually accepted cut-off, CPAP effect grows with increased use. A recent randomised study in a cohort of 3100 CPAP-treated patients, randomised in intensive versus standard interventions, has also confirmed the positive effect of a greater CPAP use (6.9 vs 5.2 h/night) on cardiovascular outcomes, indicating that a regular 5-6 hours use/night is required.

Improvement in adherence can be obtained by supportive, educational and behavioural therapy . CPAP specific education is nowadays routinely applied in the center.

Telemonitoring has also been shown to improve adherence. Other studies have added telemonitoring vs. placebo to the usual care in 45 recently diagnosed OSA patients and observed a 46% adherence improvement in the telemonitoring group after 2 months.

In another randomised trial, daily download of CPAP data and consecutive phone-call intervention to usual care in 75 OSAS patients. After 3 months, mean adherence was 321 min in the telemonitoring arm versus 207 min in the standard arm during the days of use.

T4P® is a telemonitoring unit added on CPAP device allowing to obtain a daily report of usage duration, mask leaks, pressure and apnea-hypopnea index. Data are anonymously transmitted to a secured server and analysed on a dedicated web portal.

The purpose of the present study is to assess the impact of telemonitoring on the delay to the first technical intervention after CPAP titration night in CPAP-treated OSAS patients managed in the sleep unit. The shortening of this delay could help to improve adherence during the first weeks of treatment. As secondary aim, investigators would like to assess the impact of telemonitoring on mean adherence during the first 3 months of treatment, which is a crucial period.

Material and methods Consecutive OSAS patients admitted in the sleep unit for CPAP titration night will be screened. If patients accept to participate to the study, they will be randomised between standard care or telemonitoring CPAP follow-up.

Standard care After CPAP titration night, patients are instructed to use the device each night for the whole night. They receive written instruction and can reach the sleep unit (phone call, visit) how often they need, during week days, in order to resolve any intercurrent problem interfering with their CPAP use. A group educational session for CPAP-treated patients is scheduled 1 month after and a visit to the pneumologist is scheduled 1.5 months after.

Telemonitoring follow-up In addition to standard care, the T4P® is added to the CPAP of the patient at home. Sleep lab technical staff is instructed to connect to the web portal and to analyse patient's data each Tuesdays and Fridays. In case of air leaks, persistant significant apnea-hypopnea index, use < 3h on three consecutive days, investigators have to call the patient and eventually to ask him to visit the staff of the sleep lab.

Outcomes

* delay between CPAP titration night and first intervention (phone call/visit)
* mean CPAP adherence measured during the first 3 months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with obstructive sleep apnea syndrome and AHI > 20/h, who start treatment with CPAP.

Exclusion Criteria:

* Patients already on treatment with CPAP.
* Patients leaving Belgium for more than 3 weeks during study period.
* Severe restrictive respiratory disorders.
* Severe respiratory or cardiac disease.
* Severe psychiatric disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Intervention delay (days) | 3 months
  Delay between CPAP titration night and first intervention (phone call/visit)

SECONDARY OUTCOMES:
Adherence to treatment | 3 months
  daily use of CPAP (h/day)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, Phd, Principal Investigator — CHU St. Pierre, Brussels
Locations (1):
- CHU st Pierre-sleep lab, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No